CLINICAL TRIAL: NCT04302038
Title: The Effects Potato Protein on Rates of Myofibrillar Muscle Protein Synthesis in Young Women
Acronym: APRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HIREB 4969
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Muscle Protein Synthesis
Keywords: Potato Protein; Muscle protein synthesis; Young women
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Parallel group, single blind, randomized controlled trial
Who Masked: Participant
Masking Description: Potato protein will be provided pre-mixed into prepared pudding. The control group will receive pudding without protein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potato protein (Experimental): Participants will be provided with 25 g of potato protein twice per day in addition to a diet set at the recommended daily allowance. Total protein intake for this group will be 1.6 g/kg/day
  Interventions: Dietary Supplement: Protein
- Control group (Placebo Comparator): This group will consume protein from food sources set at 0.8 /kg/day including 2 pudding placebo cups per day.
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Protein — Additional daily protein provided by potato protein.
  Arms: Potato protein
Dietary Supplement: Placebo control — No additional dietary protein (outside of 0.8 g/kg/day as provided by diet)
  Arms: Control group

SUMMARY:
This study will investigate the effects of potato protein on muscle protein synthesis over a short-term (a few hours after eating) and longer term (after two weeks of unilateral resistance exercise). Young women will be randomized to received potato protein supplementation or placebo in addition to their usual diet. Muscle biopsies will be taken and the participants will drink doubly labelled water to allow for the measurement of protein synthesis over time.

DETAILED DESCRIPTION:
The loss of skeletal muscle mass and strength with advancing age, collectively termed sarcopenia, is a primary risk factor for disability, frailty, and premature mortality. This is especially true in women, where rapid rates of decline in muscle mass and greater anabolic resistance (blunting of muscle protein synthesis [MPS] despite availability of amino acids) are experienced around the time of menopause2. Previous evidence has demonstrated that resistance exercise is an effective strategy to mitigate muscle loss in older adults, particularly in conjunction with protein supplementation. Typically, animal-based proteins are utilized in research studies; however, they may be inaccessible for older women with limited financial income or simply unattractive to the growing number of women consuming more plant-based diets. While potatoes contain lower amounts of protein compared to animal sources, the high biological value (BV~90-100) of potato protein and high consumption rates, make this food an ideal source of protein in North American diets. In fact, potatoes contribute roughly 3%-3.5% of the total daily protein intake for adults and plant-based proteins contribute 60% of dietary protein worldwide. When compared to animal sourced protein, potatoes are readily available and are a highly sustainable food source. Consequently, potatoes represent an accessible, cost-effective protein source for the growing aging population. However, the efficacy of a diet rich in potato protein to stimulate an increase in integrated rates of MPS, which are the basis for muscle growth, in women has not been investigated. Therefore, while the eventual target consumer will be all women, young and old, firstly we will demonstrate the effectiveness of potato based protein to stimulate MPS in young women.

Twenty-four healthy young women (18-29 yrs) will be recruited to participate in this parallel group, double blind, randomized controlled trial. Participants will be randomized to either supplementary isolated potato protein and unilateral resistance training, or unilateral resistance training alone as placebo (with usual dietary practices, protein clamped at 0.8 g/kg/day). Participants will engage in unilateral resistance training 3 times per wk for 2 wk. To assess the anabolic properties of potato protein, the women in the potato protein group will ingest 25 g of isolated potato protein 2 times a day. On the day of resistance exercise one serving will be provided immediately after the cessation of training. The placebo group will follow the same supplement schedule, but with a placebo. Integrated rates of myofibrillar MPS will be assessed with the precursor-product method using deuterium labeled water (70% D2O).

ELIGIBILITY:
Inclusion Criteria:

* meet the age requirements
* Female sex

Exclusion Criteria:

* Significant loss or gain of body mass in the past 6 months (>2 kg)
* Regular use of: non-steroidal anti-inflammatory drugs
* History of chronic disease
* Current or recently active or remised cancer
* Infectious disease; and/or gastrointestinal disease
* Consuming a vegetarian or vegan diet = Any condition or injury that would preclude them from participating in resistance exercise

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 17 days
  Myofibrillar protein synthesis via measurement of deuterated (doubly) labeled water

SECONDARY OUTCOMES:
Protein expression | 17 days
  Western blot analysis to determine total protein expression of the proteins involved in the muscle protein synthesis pathway

CONTACTS AND LOCATIONS:
Locations (1):
- Ivor Wynne Centre, Hamilton, Ca-on, Canada

IPD SHARING:
Plan to Share IPD: No